CLINICAL TRIAL: NCT00820261
Title: Molecular Epidemiology of Rotavirus Diarrhea Among Infants and Young Children Attending Maua Methodist Hospital, Kenya
Acronym: Rotavirus
Status: Completed | Type: Observational
Sponsor: Institute of Primate Research (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Atunga Nyachieo, Senior Research Scientist, Institute of Primate Research
Other Study IDs: IISP35341; IISP35341
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Rotavirus
Keywords: Genotypes; Epidemiology; Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Fluid Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The positive samples will be evaluated by sodium dodecyl polyacrylamide gel electrophoresis (SDS-PAGE) to determine the electropherotypes and genotyped using reverse transcriptase polymerase chain reaction (RT-PCR) on VP7 and VP4 gene and sequencing. Also, these positive samples will be retained for quality assurance and quality control.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diarrhea: children and infants (less than 5 years of age) presenting with severe diarrhea will be enrolled
  Interventions: Other: oral rehydration therapy for diarrhea cases

INTERVENTIONS:
Other: oral rehydration therapy for diarrhea cases — Since rotavirus infection is a viral infection with no drug remedy, diarrhea cases will be managed according to the standard WHO protocol for the management of diarrhea. This will include oral rehydration treatment.

SUMMARY:
Rotavirus is the most common cause of severe infantile diarrhoea disease in infants and young children below five years worldwide. It is associated with high cases of morbidity and mortality and it is estimated that up to 600,000 deaths in young children occur annually in the less developed countries and approximately 150,000-200,000 deaths occur in Africa alone. In Kenya, most rotavirus surveillance work has been done in Nairobi (an urban setting). Other parts e.g eastern Kenya, limited data is available and hence the prevalence and burden of rotavirus disease is under-estimated. We therefore hypothesize that rotavirus prevalence is high in Meru,Maua (a rural setting)and hence we designed a study to evaluate this.

This is a prospective study to determine, the rotavirus disease burden and epidemiology in infants and children with severe diarrhoea hospitalized in three sentinel hospital in the eastern part of Kenya (Maua Methodist hospital) will be carried out during the period January 2009 to December 2010.

Faecal samples will be collected from infants and children admitted with acute diarrhoea and screened first for the presence of human serotype A rotavirus antigen using commercially available enzyme linked immunosorbent assay kit (ELISA).

The positive samples will be evaluated by sodium dodecyl polyacrylamide gel electrophoresis (SDS-PAGE) to determine the electropherotypes and genotyped using reverse transcriptase polymerase chain reaction (RT-PCR) on VP7 and VP4 gene.

These data/ results generated from this project will add crucial information on the rotavirus strains circulating in the eastern part of Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Only children under 5 years of age who present with acute diarrhea having experienced an episode of 3 looser than normal or watery stools in a 24-hour period with or without episodes of vomiting will be enrolled in this study.
* And the diarrhea should last for ≤ 7 days.
* Clinical studies have indicated that the incubation period for rotavirus illness is less than 48hrs and usually will last for 5-7days (Steele, 1998) Based on this fact, and as per the WHO's Generic Protocol for Hospital based Surveillance of Rotavirus Gastroenteritis in children under 5 years of age (WHO Generic protocol, 2002)

Exclusion Criteria:

* Children more than 5 years of age and with diarrhea lasting > 7 seven days and having bloody diarrhea will be excluded in the study.
* This is as per the who's generic protocol for hospital based surveillance of rotavirus gastroenteritis in children under 5 years of age (WHO Generic Protocol, 2002)

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Stool specimens will be collected from infants and young children below 5 years of age with severe diarrhea hospitalized in two government hospital (Maua Methodist hospital, during a two (2) year period
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2009-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percentage prevalence of rotavirus positive cases | 3 years

SECONDARY OUTCOMES:
Any novel rotavirus strain detected by sequencing | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Atunga Nyachieo, PhD Biomedical Sciences, Principal Investigator — Institute of Primate Research, Kenya; Nicholas M Kiulia, BSc Med Micro, Study Director — Institute of Primate Research, Kenya; Maureen B Taylor, DSc Virology, Principal Investigator — Medical Virology Department, Univesity of Pretoria, South Africa; Walda van Zyl, PhD Virology, Principal Investigator — Medical Virology Department, Univesity of Pretoria, South Africa
Locations (1):
- Maua Methodist Hospital, Maua, Eastern, Kenya